CLINICAL TRIAL: NCT03928574
Title: Ultrasound-Guided Plane Versus Conventional Block of the Medial Brachial Cutaneous and the Intercostobrachial Nerves：A Retrospective Observational Study
Brief Title: USG Block of Cutaneous Nerves of the Arm
Status: Completed | Type: Observational
Sponsor: Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019CZTCWM1
Record Dates: First submitted 2018-05-08; First posted 2019-04-26 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2019-04

CONDITIONS: Nerve Block
Keywords: Ultrasound-Guided Plane Block; Conventional Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound-Guided: Ultrasound-Guided Plane Block
  Interventions: Procedure: Ultrasound-Guided Plane Block
- Conventional: Conventional Block
  Interventions: Procedure: Conventional Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Plane Block — Ultrasound-Guided Plane Block Medial Brachial Cutaneous and the Intercostobrachial Nerves
  Groups: Ultrasound-Guided
Procedure: Conventional Block — Conventional Block Medial Brachial Cutaneous and the Intercostobrachial Nerves
  Groups: Conventional

SUMMARY:
For superficial surgery of anteromedial and posteromedial surfaces of the upper arm, the medial brachial cutaneous nerve (MBCN) and the intercostobrachial nerve (ICBN) must be selectively blocked, in addition to an axillary brachial plexus block. We compared efficacy of ultrasound-guided (USG) versus conventional block of the MBCN and the ICBN.

DETAILED DESCRIPTION:
The primary objective of our study was to compare the effectiveness of conventional and USG blocks of the MBCN and the ICBN in the axillary fossa. Our hypothesis was that the proportion of patients with complete anesthesia in the entire posteromedial and anteromedial surface of the arm would be greater if a USG technique were used, compared with a conventional technique. The secondary objectives were onset time of complete anesthesia, volume of local anesthetic used for the procedure, tourniquet tolerance during surgery, and ultrasound visibility of MBCN and ICBN.

ELIGIBILITY:
Inclusion Criteria:

* Surgery of the distal upper limb : hand, forearm, lower third of the arm ,including the elbow
* Urgent or planned surgery
* Locoregional anesthesia : axillary brachial plexus block, completed by a medial brachial cutaneous nerve block and an intercostobrachial nerve block

Exclusion Criteria:

* Refused to sign informed consent
* Pregnant women
* Allergic to the local anesthetic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete anesthesia | At time 20 minutes after the medial brachial cutaneous nerve and the intercostobrachial nerve block
  Number of participants with complete anesthesia of the arm in region innervated by the MBCN and the ICBN

SECONDARY OUTCOMES:
Number of participants with complete anesthesia, with reduced sensitivity and with absence of anesthesia | At times 5, 10, 15, 20 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
  Number of participants with complete anesthesia, with reduced sensitivity and with absence of anesthesia at times 5, 10, 15, 20 minutes (except primary outcome) in the areas of the medial brachial cutaneous nerve and the intercostobrachial nerve
Volume of local anesthetic | After nerve block immediately
  The volume (in milliliters) of 1% lidocaine used for the medial brachial cutaneous nerve and the intercostobrachial nerve block
Tourniquet tolerance | 3 hours after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
  Number of patients with comfortable feeling, with unpleasant sensations and with pains during surgery, in the areas of the medial brachial cutaneous nerve and the intercostobrachial nerve
Good ultrasound view of theses nerves before and after the injection of the local anesthetic | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
  Number of participants (of the ultrasound-guided group) with good ultrasound view of theses nerves before and after the injection of the local anesthetic
Bad ultrasound view of theses nerves before the injection and good ultrasound view of theses nerves after the injection of the local anesthetic | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
  Number of participants (of the ultrasound-guided group) with bad ultrasound view of theses nerves before the injection and good ultrasound view of theses nerves after the injection of the local anesthetic
Bad ultrasound view of theses nerves before and after the injection of the local anesthetic | 5 minutes after the achievement of the medial brachial cutaneous nerve block and the intercostobrachial nerve block
  Number of participants (of the ultrasound-guided group) with bad ultrasound view of theses nerves before and after the injection of the local anesthetic

CONTACTS AND LOCATIONS:
Overall Officials: Ruizha Lv, M.D, Principal Investigator — Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided